CLINICAL TRIAL: NCT04183322
Title: Reactogenicity and Immunogenicity of Pneumococcal Conjugate Vaccination in Non-pregnant Papua New Guinean Women
Brief Title: PCV13 in Non-pregnant Papua New Guinean Women
Status: Completed | Type: Observational
Sponsor: Telethon Kids Institute (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB 1515
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal conjugate vaccine; PCV; Reactogenicity; Immunogenicity; Women childbearing age
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women of childbearing age: Healthy non-pregnant women between 18 and 45 years old living in Goroka, Papua New Guinea, will receive one dose of 13-valent pneumococcal conjugate vaccine (PCV).
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine
  Other Names: PCV13; 13-valent PCV; Prevnar13; Prevenar13

SUMMARY:
This is an observational study to determine the reactogenicity and immunogenicity of pneumococcal conjugate vaccine in non-pregnant women of reproductive age in Papua New Guinea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-pregnant
* 18-45 years old

Exclusion Criteria:

* Known hypersensitivity to any vaccine component
* Known/suspected to be immunocompromised
* Receipt of corticosteroids ≤30 days before
* Pregnant (pregnancy tests will be performed)
* Not being well at the time of vaccination
* Plan to travel out of the area in the month post-vaccination

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: 50 healthy non-pregnant women aged between 18-45 years old living in Goroka, Papua New Guinea.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 28 days
  Mean Fold Increase (MFI; and 95% CI) in vaccine-serotype specific IgG concentrations at 28 days after compared to baseline (before vaccination)

SECONDARY OUTCOMES:
Reactogenicity | 24-48 hours after vaccination
  Proportion (% & 95% CI) of participants with local and systemic side effects 24-48 hours after vaccination
Adverse events | 28 days
  Proportion (% & 95% CI) of participants reporting any unexpected adverse effect (AE) during 28 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Papua New Guinea Institute of Medical Research, Goroka, Eastern Hghlands Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javati S, Masiria G, Elizah A, Matlam JP, Ford R, Richmond PC, Lehmann D, Pomat WS, van den Biggelaar AHJ. An observational study of the reactogenicity and immunogenicity of 13-valent pneumococcal conjugate vaccine in women of childbearing age in Papua New Guinea. Pneumonia (Nathan). 2020 Nov 25;12(1):13. doi: 10.1186/s41479-020-00076-1. PMID 33292822